CLINICAL TRIAL: NCT03291600
Title: Virtual Psychiatric Care for Perinatal Depression (Virtual-PND): A Pilot Randomized Controlled Trial
Brief Title: Virtual Psychiatric Care for Perinatal Depression
Acronym: Virtual-PND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Women's College Hospital (Other)
Collaborators: Sinai Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20170061B
Record Dates: First submitted 2017-09-19; First posted 2017-09-25 (Actual); Last update posted 2019-02-05 (Actual); Status verified 2019-02

CONDITIONS: Perinatal Depression

STUDY DESIGN:
Intervention Model Description: Behavioral: Virtual Psychiatric Care for Perinatal Depression
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual Psychiatric Care Group (Experimental): Participants randomized to the intervention group will have the option to receive video-based psychiatrist care in addition to care as usual. Participants will be assigned to begin immediately after randomization.
  Interventions: Behavioral: Virtual Psychiatric Care
- Control Group (No Intervention): Women allocated to the control condition will receive care as usual (in-person psychiatric care) from the study site to which they were referred.

INTERVENTIONS:
Behavioral: Virtual Psychiatric Care — Virtual psychiatric care for perinatal depression will be offered to participants, in addition to care as usual, for a 12-week period by their treating perinatal psychiatrist. Virtual care will be delivered by video-based visits through the Ontario Telemedicine Network (OTN). The treating psychiatrist may request that an intervention group participant present for in-person care at any visit, and this may include need for behavioural activation, or another health-related indication at the discretion of the treating psychiatrist.
  Arms: Virtual Psychiatric Care Group

SUMMARY:
Perinatal depression occurs in 15% of pregnant women and new mothers, yet as few as 1 in 5 receive adequate treatment. It has a negative impact on the woman herself, as well as a potential for serious consequences for her child. Virtual psychiatric care is a potential model that may provide accessible mental health care during this time, as barriers to in-person care often include unpredictable infant schedules, competing childcare demands, or travel/cost challenges. The Virtual-PND intervention consists of 12-weeks of the option of supplementing in-person psychiatric care with secure, in-home real-time video-visits through the Ontario Telemedicine Network. This pilot RCT will demonstrate the feasibility of proceeding to a future large-scale RCT evaluation of virtual psychiatric care for this population.

DETAILED DESCRIPTION:
This is a two-site pilot randomized controlled trial (RCT) to evaluate the feasibility of a Virtual Psychiatric Care for Perinatal Depression (Virtual-PND) intervention protocol, comparing virtual care to in-person care only. Participants will be pregnant or postpartum women with a major depressive disorder who are referred for care at one of the participating study sites. Each study site is a specialist reproductive psychiatric program where women from the greater Toronto area are referred, and generally treated with in-person care. Those randomized to the virtual care group will be able to receive psychiatric visits with video-based visits. Those randomized to the in-person care group will receive in-person care only, as per usual clinical practice at the study sites. The length of the active treatment phase will be 12 weeks from enrolment. The overall objective of this pilot RCT is to determine the feasibility of conducting a larger RCT to evaluate the efficacy of the treatment model, comparing outcomes among those with and without access to virtual care, and cost-effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* Pregnant or 0-12 months postpartum
* Experiencing clinically significant depressive symptoms (defined as a score of ≥12 on the Edinburgh Postnatal Depressive Scale, EPDS, during eligibility screening)
* Able to access the internet on a device (i.e. mobile phone, tablet, personal computer) with video-visit capacity (including web camera and speakers)
* Comfortable with email communication

Exclusion Criteria:

* Active alcohol/substance use disorder in the past 12 months
* Active suicidal ideation
* Current mania or psychosis
* Unsuitable for virtual care, as per assessment of the treating psychiatrist

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2017-10-24 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Recruitment Feasibility (Recruitment Feasibility) | One year from when the study starts enrolling participants
  The number of women recruited to the study at each site

SECONDARY OUTCOMES:
Edinburgh Postnatal Depressive Scale (EPDS) | At 12 weeks post-randomization
  The investigators will measure depressive symptoms using the EPDS, a self-report, 10-item depression screening measure that has been validated for use in pregnancy. EPDS scores >12 are predictive of a diagnosis of major depressive disorder.
State-Trait Anxiety Inventory (STAI) | At 12 weeks post-randomization
  The investigators will measure anxious symptoms using the STAI, a self-report, 40-item anxiety screening measure that has shown good discriminate validity in perinatal populations. STAI scores >48 are predictive of having an anxiety disorder diagnosis.
Parenting Stress Index, Short Form (PSI) | At 12 weeks post-randomization
  The investigators will measure stress in the parent-child relationship using the PSI short form, a 36-item measure which consists of three sub-scales.
Recruitment Feasibility (Recruitment Eligibility) | One year from when the study starts enrolling participants
  The proportion of participants eligible to participate at each recruitment site
Recruitment Feasibility (Enrollment) | From enrollment to first treatment visit
  Average length of time from enrollment to 1st psychiatrist visit
Intervention Acceptability (Qualitative - participants) | At 12 weeks post-randomization
  Virtual-PND Participant Program Evaluation Questionnaire. This is comprised of Likert-type scale questions to elicit feedback on acceptability of the virtual care experience and model.
Intervention Acceptability (Qualitative - physicians) | At 12 weeks post-randomization
  Virtual-PND Physician Program Evaluation Questionnaire. This is comprised of open and closed-ended questions to elicit feedback on the acceptability of the virtual care experience and model.
Intervention Acceptability (Patient-Reported Costs) | At 12 weeks post-randomization
  Patient-Reported Costs Questionnaire. This is comprised of open and closed-ended questions regarding: a) time spent travelling to visits and on missed work; and b) cost of travel, food, childcare and data charges.
Intervention Acceptability (Clinical visits) | Between randomization and 12 weeks post-randomization
  Medical chart review - number of psychiatrist visits (overall, in person, and virtual), and number of minutes per visit.
Trial Protocol Adherence (Study Measure Completion) | At 12 weeks post-randomization
  Proportion of participants who complete follow-up measures.

CONTACTS AND LOCATIONS:
Overall Officials: Lori Wasserman, MD, FRCPC, Principal Investigator — Women's College Hospital; Ariel Dalfen, MD, FRCPC, Principal Investigator — Sinai Health System
Locations (2):
- Canada (2):
  - Mount Sinai Hospital, Toronto, Ontario
  - Women's College Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No